CLINICAL TRIAL: NCT05038137
Title: The Effects of Time Restricted Feeding on AGE-RAGE Signaling in Women at High Risk for Breast Cancer
Brief Title: Time Restricted Eating on Cancer Risk
Acronym: TREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109489
Record Dates: First submitted 2021-08-31; First posted 2021-09-08 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Pre-diabetes; Breast Cancer; Time Restricted Feeding
MeSH Terms: conditions — Glucose Intolerance; Breast Neoplasms; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: Visit 1 at 0 weeks, followed by 2 week run-in and then randomization. Visit 2 at 14 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time restricted feeding (Experimental): daily eating period of 8 hours, before 8 PM for 12 weeks
  Interventions: Behavioral: Time restricted feeding
- Control (Active Comparator): daily eating period ≥ 12 hours for 12 weeks
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Time restricted feeding — Participants will eat all food during a self selected 8 hour eating window prior to 8:00 PM.
  Arms: Time restricted feeding
Behavioral: Control — Participants will have a daily eating period equal to or greater than 12 hours.
  Arms: Control

SUMMARY:
Participants will be randomly assigned to either the time restricted feeding group with a daily eating period of 8 hours or the control group with a daily eating period of greater than or equal to 12 hours. There are 2 in-person study visits to have blood, urine and vital signs collected and 8 remote or phone visits with a psychologist or dietician to assist with the eating schedule. The study will take last 3 1/2 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 40 and ≤ 67;
* Postmenopausal women (no menstrual periods in the preceding 12 or more months) with pre-diabetes (A1C 5.7-6.4% and/or fasting glucose 100-125 mg/dL). A1c lab and/or fasting glucose criteria will need to be met within 12 months of signing consent form, can be obtained from prior lab result or study prescreening testing;
* Own a smart phone with internet connection and capable of receiving and sending text messages and taking photographs;

Exclusion Criteria:

* Tobacco use (current or within last 2 years);
* Active malignancy or history of cancer;
* History of known liver disease (by serology: aspartate aminotransferase or alanine aminotransferase ≥ 3 times above upper limit of normal determined by lab review, imaging or biopsy: determined by patient history);
* History of kidney disease (patient history and/or estimated glomerular filtration rate less than 45 mL/min/1.73m²);
* History of diabetes mellitus:
* History of cardiovascular disease (MI, CHF);
* Current prescription medication use for diabetes;
* Medication affecting glucose metabolism or appetite or immunosuppression;
* Dietary restrictions: currently following vegetarian or vegan dietary pattern;
* Currently following intermittent fasting or time restricted feeding pattern or use in the last 3 months;
* Night shift worker (work schedule does not involve any period of work from 10 PM to 5 AM either on a regular or rotating basis);
* History of weight loss >5% in the last 3 months;
* History of weight loss surgery.
* BMI≥40 kg/m² exclusion;
* After informed consent and run in period: Insufficient documented food photography/annotated entries (does not log at least two entries a day for 10 of 14 days) during run in period will be excluded from randomization in to the intervention period.

Ages: 40 Years to 67 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal women (no menstrual periods in the preceding 12 or more months) with pre-diabetes (A1C 5.7-6.4% and/or fasting glucose 100-125 mg/dL).
Enrollment: 29 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harsha Karanchi, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Time Restricted Feeding: daily eating period of 8 hours, before 8 PM
  Time restricted feeding: Participants will eat all food during a self selected 8 hour eating window prior to 8:00 PM for 12 weeks.
- Control: daily eating period ≥ 12 hours
  Control: Participants will have a daily eating period equal to or greater than 12 hours for 12 weeks.
Period: Overall Study
Arm/Group | Time Restricted Feeding | Control
Started | 15 | 14
Completed | 15 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Time Restricted Feeding: daily eating period of 8 hours, before 8 PM
  Time restricted feeding: Participants will eat all food during a self selected 8 hour eating window prior to 8:00 PM.
- Control: daily eating period ≥ 12 hours
  Control: Participants will have a daily eating period equal to or greater than 12 hours.
- Total: Total of all reporting groups
Arm/Group | Time Restricted Feeding | Control | Total
Number analyzed (Participants) | 15 | 14 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.4 (6.0) | 58.5 (6.1) | 58.4 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 10 | 8 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 15 | 14 | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Advanced Glycation End Products (AGE) as Assessed by Plasma
Description: Estimated mean levels within the intervention and the control groups of the study. Effect size will be estimated via 95% confidence intervals within and between groups.
Time Frame: Visit 1 (0 weeks), Visit 2 (14 weeks)
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 15 | 14
ng/mL
  Visit 1 (0 weeks) | 5.82 [5.49 to 6.15] | 6.38 [5.71 to 7.05]
  Visit 2 (14 weeks) | 5.82 [5.45 to 6.20] | 6.40 [5.88 to 6.93]

2. Primary Outcome: Change in sRAGE(Soluble Receptor for AGE) Levels
Description: Estimated mean levels within the intervention and the control groups of the study. Effect size will estimated via 95% confidence intervals within and between groups.
Time Frame: Visit 1 (0 weeks), Visit 2 (14 weeks)
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 15 | 14
ng/mL
  Visit 1 (0 weeks) | 2.77 [2.63 to 2.90] | 2.65 [2.51 to 2.79]
  Visit 2 (14 weeks) | 2.64 [2.47 to 2.80] | 2.58 [2.42 to 2.75]

3. Primary Outcome: Assess Feasibility and Adherence to Time Period of Eating Recommendations in Both Study Groups.
Description: Percentage of dietary visits that participant reported compliance with randomized eating period.
Time Frame: Visit 1 (0 weeks), Visit 2 (14 weeks)
Measure: Mean (Full Range); unit: Percentage of visits
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 15 | 14
Percentage of visits | 90.1 [0 to 100] | 83.3 [14.3 to 100]

4. Secondary Outcome: Change in Fasting Insulin-like Growth Factor-1 (IGF-1) Levels
Description: as for outcome 1
Time Frame: Visit 1 (0 weeks), Visit 2 (14 weeks)
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 15 | 14
ng/ml | 2.5 (24) | .01 (16)

5. Secondary Outcome: Change in Fasting Insulin Levels
Description: as for outcome 1
Time Frame: Visit 1 (0 weeks), Visit 2 (14 weeks)
Measure: Mean (95% Confidence Interval); unit: µU/ml
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 15 | 14
µU/ml | -0.6 [-9.3 to 2.7] | 1.0 [0.3 to 5.3]

6. Secondary Outcome: Difference in Glasgow Prognostic Scoring System
Description: The Glasgow Prognostic Score (GPS) reflects systemic inflammatory process. GPS is a three-tiered score [0: normal C-reactive protein (CRP) and albumin; 1: one abnormal result; 2: increased CRP and low albumin]. Higher score means worse outcome.
Time Frame: Visit 1 (0 weeks), Visit 2 (14 weeks)
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 15 | 14
score on a scale | 0 [0 to 0] | 0 [0 to 0]

7. Secondary Outcome: Change in 24 Hour Urinary AGE Levels
Description: Estimated mean levels within the intervention and the control groups of the study. Effect size will be estimated by the 95% confidence intervals within and between groups.
Time Frame: Visit 1 (0 weeks), Visit 2 (14 weeks)
Measure: Mean (95% Confidence Interval); unit: ng/mL
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 15 | 14
ng/mL
  Visit 1 (0 weeks) | 6.51 [6.10 to 6.92] | 6.69 [6.18 to 7.20]
  Visit 2 (14 weeks) | 5.82 [5.33 to 6.31] | 6.02 [5.55 to 6.49]

8. Secondary Outcome: Adherence to Virtual Visit With Psychologist or Dietician
Description: Percentage of expected visits attended.
Time Frame: Visit 1 (0 weeks), Visit 2 (14 weeks)
Measure: Mean (Full Range); unit: Percentage
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 15 | 14
Percentage | 97.5 [75 to 100] | 98.2 [87.5 to 100]

9. Secondary Outcome: Adherence to Time Period of Eating Recommendation in Both Study Groups: Self Reporting During Virtual Visits and Through Food Photography / Annotated Entries.
Description: Proportion of dietary visits where participants reported compliance with randomized eating period, assessed through self-report during virtual visits and via food photography/annotated entries.
Time Frame: Visit 1 (0 weeks), Visit 2 (14 weeks)
Reporting Status: Not Posted, anticipated posting 2026-06

10. Secondary Outcome: Percentage of Participants With Stable Chronotype Between Baseline and End of Study
Description: Stability in chronotype (normal, delayed, or advanced) was assessed using 2-week sleep diaries at baseline and end of study. Stability was defined as no change in chronotype classification between Visit 1 and Visit 2.
Time Frame: Visit 1 (0 weeks), Visit 2 (14 weeks)
Population: All randomized participants who completed both baseline and end-of-study sleep diaries were included in the analysis. Stability was defined as no change in chronotype classification between Visit 1 and Visit 2.
Measure: Number (95% Confidence Interval); unit: % of participants with stable chronotype
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 13 | 14
% of participants with stable chronotype | 0.923 [0.655 to 0.992] | 0.857 [0.603 to 0.960]

11. Secondary Outcome: Mean Glucose at Visit 2
Description: Mean glucose level calculated as the average of continuous glucose monitoring (CGM) data collected during the final 14 days of the intervention period (Visit 2).
Time Frame: Final 14 days of intervention period (Visit 2).
Population: All randomized participants who completed CGM monitoring during the final 14 days of the intervention period were included in the analysis. Mean glucose was calculated as the average of all CGM readings during this period.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 13 | 11
mg/dL | 113.8 [108.8 to 118.8] | 101.9 [96 to 107.8]

12. Secondary Outcome: Glucose Management Indicator (GMI) at Visit 2
Description: GMI percentage derived from CGM data collected during the final 14 days of the intervention period (Visit 2).
Time Frame: Visit 2 (14 weeks)
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 13 | 11
percentage | 6 [5.9 to 6.2] | 5.8 [5.6 to 5.9]

13. Secondary Outcome: Glucose Variability at Visit 2
Description: Coefficient of variation of glucose levels derived from CGM data during the final 14 days of the intervention period (Visit 2).
Time Frame: Visit 2 (14 weeks)
Measure: Mean (95% Confidence Interval); unit: percentage
Arm/Group | Time Restricted Feeding | Control
Number analyzed (Participants) | 13 | 11
percentage | 18 [16 to 20] | 17.6 [14.8 to 20.5]

ADVERSE EVENTS:
Time Frame: 14 weeks
Arm/Group | Time Restricted Feeding | Control
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/14
Other Adverse Events (participants affected / at risk) | 0/15 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/37/NCT05038137/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/37/NCT05038137/ICF_000.pdf